CLINICAL TRIAL: NCT06701773
Title: Computational Fluid Dynamics Predicting Intraprosthetic Thrombus Formation and Progression Following Endovascular Aortic Repair: a Two-center Retrospective Study
Brief Title: Computational Fluid Dynamics Predicting Intraprosthetic Thrombus Formation and Progression Following EVAR
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Wei Wang, Professor, Xiangya Hospital of Central South University
Other Study IDs: 2024030373
Record Dates: First submitted 2024-11-17; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Intraprosthetic Thrombus; Limb Graft Occlusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intraprosthetic thrombus Group: presence of intraprosthetic thrombus according to the postoperative CTA
- Non-intraprosthetic thrombus Group: absence of intraprosthetic thrombus according to the postoperative CTA

SUMMARY:
Intraprosthetic thrombus (IPT) formation and its progression to limb graft occlusion (LGO) are significant complications following endovascular aneurysm repair (EVAR). Morphological metrics based on preoperative CTA have limited predictive value for these complications. This study aims to assess the potential of computational fluid dynamics (CFD) in predicting IPT formation and its progression to LGO after EVAR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above;
2. Patients undergone endovascular aneurysm repair;
3. Signed informed consent forms, willing to receive treatments.

Exclusion Criteria:

1. inflammatory aortic aneurysm;
2. patients diagnosed with connective tissue diseases;
3. patients diagnosed with atrial fibrillation;
4. patients lacking post-operative CTA;
5. Patients who are participating in other clinical projects;
6. Patients are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergone endovascular aneurysm repair.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Degree of intraprosthetic thrombus in limb graft | From January 2014 to June 2024
  Evaluate the area of thrombus occupying the lumen using postoperative CTA

SECONDARY OUTCOMES:
Disease-related complications | From January 2014 to June 2024
  Disease-related complications associated with intraprosthetic thrombus or limb graft occlusion, such as thromboembolic events